CLINICAL TRIAL: NCT06641687
Title: Oral Sucrose for Pain Management During Flexible Nasolaryngoscopy
Brief Title: Be Sweet to Babies During Nasolaryngoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Nikolaus Wolter, Staff Otolaryngologist, Department of Otolaryngology - Head & Neck Surgery, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000081486
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Infant Conditions
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sterile water (Placebo Comparator): Participants will be given sterile water which does not contain sugar and is used as a placebo
  Interventions: Other: Sterile water
- Sucrose solution (Experimental): Participants will be given sugar water which contains 24% sucrose. As per pharmacy at The Hospital for Sick Children, Sucrose is not classified as a drug as per Health Canada.
  Interventions: Other: 24% Sucrose

INTERVENTIONS:
Other: 24% Sucrose — Participants will be given either sugar water (24% sucrose) randomly
  Arms: Sucrose solution
Other: Sterile water — Participants will be given sterile water randomly
  Arms: Sterile water

SUMMARY:
The investigators want to know if sugar water containing 24% sucrose is helpful in reducing pain in babies during scopes.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of oral sucrose on pain or distress in outpatient infants undergoing flexible nasolaryngoscopy during a scheduled appointment at the SickKids Pediatric Otolaryngology Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patient <12 months of age;
* Scheduled for an appointment with Dr. Nikolaus Wolter or Dr. Jennifer Siu, who are Staff Pediatric Otolaryngologists at the Hospital for Sick Children, or Meghan Tepsich, a complex airway Nurse Practitioner at SickKids;
* Requiring flexible nasolaryngoscopy for diagnostic purposes;
* Accompanied by caregivers who provided consent.

Exclusion Criteria:

* Patient >12 months of age
* Infants <37 weeks corrected gestational age
* Infants with decreased level of consciousness or delayed neuromuscular development with limited pain response
* Infants who have received acute/urgent /emergent airway assessment such as respiratory distress or a foreign body, etc.
* Infants who have received topical anesthesia (topical decongestant/anesthetic spray)
* Infants with the following conditions, where oral sucrose is contraindicated or ineffective:

  * Carbohydrate intolerance
  * Decreased level of consciousness or heavy sedation
  * Absent gag reflex
  * Non-functional gastrointestinal tract
  * History of aspiration, tracheoesophageal fistula
  * Necrotizing enterocolitis
* Infants whose parents did not consent to enrolling their child in the study, including randomization into either arm of the study due to preference for a given intervention
* Any other circumstance in which consent for participation in the study was not obtained prior to the scope

Infants will also be excluded from the study if they present with conditions in which FNL is contraindicated:

* Severe respiratory distress
* Post-palliative systemic artery to pulmonary artery shunt
* Single ventricle congenital heart disease

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | up to 7 months
  Clinical pain scores change after flexible nasolaryngoscopy (FNL) in 60 infants under 12 months of age following the use of sucrose solutions. The EVENDOL scale is a validated 15-point scale (range of 0-15) developed for children with presenting, prolonged, or procedural pain. Infant pain observations are ranked from 0-3 based on 5 different observations: (1) vocal or verbal expression, (2) facial expression, (3) movements, (4) postures, and (5) interactions with the environment. Higher scores mean a worse outcome (more pain).

SECONDARY OUTCOMES:
Crying time | up to 7 months
  Crying time (second - s) after FNL in 60 infants under 12 months of age following the use of oral sucrose solutions.
Maximum Heart rate | up to 7 months
  Maximum heart rate (beats per minute - bpm) as measured by a pulse oximeter during FNL in 60 infants under 12 months of age following the use of oral sucrose solutions.
Time to baseline | up to 7 months
  The time taken for heart rate to return to baseline (second - s) as measured by a pulse oximeter during FNL in 60 infants under 12 months of age following the use of oral sucrose solutions.
Plantar skin conductance | up to 7 months
  Plantar skin conductance (μS) during FNL in 60 infants under 12 months of age as measured by maximum peaks per second, following the use of oral sucrose solutions.
Duration of clinic visit | up to 7 months
  Duration of clinic visits (minutes) following the administration of oral sucrose.
Caregiver impression | up to 7 months
  Caregiver impression of infant discomfort following the use of oral sucrose based on Wong-Baker FACES Pain Rating Scale (range of 0-10), higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus E. Wolter, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We are not going to make individual patient data available to others.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT06641687/Prot_SAP_000.pdf